CLINICAL TRIAL: NCT03572647
Title: Randomized Clinical Study for Pharmacokinetics and Pharmacodynamics Assessment of Drug Eritromax, Marketed by the Blausiegel Laboratory, Compared to Drug Eprex, Produced by Janssen-Cilag Laboratory, in Healthy Subjects.
Brief Title: Pharmacokinetics and Pharmacodynamics Assessment of Drug Eritromax Compared to Eprex in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Collaborators: Blau Farmaceutica S.A. (Industry)
Responsible Party: Principal Investigator, Azidus Brasil, Principal Investigator Alexandre Frederico, Azidus Brasil
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EPOBLA0711I
Record Dates: First submitted 2011-11-03; First posted 2018-06-28 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Renal Insufficiency, Chronic
Keywords: Erythropoeitin; Chronic kidney disease; Anaemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test ERITROMAX (Experimental): Blausiegel Industria e Comercio Ltda. Recombinant Human Erythropoietin (ERITROMAX)
  Interventions: Drug: Eritromax
- EPREX (Active Comparator): Janssen-Cilag Recombinant Human Erythropoietin (EPREX)
  Interventions: Drug: Eprex

INTERVENTIONS:
Drug: Eritromax — The subjects will receive a single dose of 4000 IU epoetin alfa in each period, according to randomisation.
  Other Names: epoetin alfa
  Arms: Test ERITROMAX
Drug: Eprex — The subjects will receive a single dose of 4000 IU epoetin alfa in each period, according to randomisation.
  Other Names: epoetin alfa
  Arms: EPREX

SUMMARY:
The epoetin is a glycoprotein and endogenous hormone, which is primarily synthesized by specific epithelial cells lining the kidney peritubular capillaries, and regulates continuous formation of red blood cells. This is a pharmacokinetics and pharmacodynamics study, in which each subject will receive the investigational product in different periods, as randomisation (Teste or Comparator). The evaluation of the profile included serum dosage of medications and reticulocyte count in peripheral blood.

DETAILED DESCRIPTION:
This a prospective randomized and crossover study for evaluation of pharmacokinetics and pharmacodynamics of two epoetins formulations. The subjects will receive in each confinement period 4000 IU one of the investigational product subcutaneously, according to randomisation, separated by a washout period of 4 weeks. The evaluation of the profile between products included serum dosage of medications and reticulocyte count in peripheral blood. Safety evaluation data will include report od all adverse events (including type, frequency, intensity, seriousness, severity and action taken related to the investigational product study).

ELIGIBILITY:
Inclusion Criteria:

* Confirm the voluntary participation and agree to all the purposes of the study by signing and dating the IC in two ways;
* Being male, aged between 20 and 55 years, clinically healthy;
* BMI between 18 and 25;
* Results of examination of hemoglobin between 13.8 and 15.4 g / dL and hematocrit between 41% and 49%;
* Results of VCM, HBMC, platelets and leukocytes within the normal range:

VCM = Between 82 to 98. Among the HBMC = 26 to 34. Among the platelets = 150,000 to 400,000 units per mL. Among the WBC = 3,500 to 10,500 units per mL and without cellular atypia.

* Serum ferritin = Male between 36 to 262 mcg / L and women between 24 to 155 mcg / L;
* Reticulocyte count in peripheral blood ≤ 3%;
* Serum erythropoietin less than 30 mIU / mL.

Exclusion Criteria:

* Participation in clinical trials in the 12 months preceding the survey;
* Presence of iron deficiency anemia;
* Presence of pulmonary diseases, cardiovascular, neurological, endocrine, gastrointestinal, genitourinary or other systems;
* Acute disease in the period of 07 days prior to inclusion;
* Chronic administration of medication to determine, such as high blood pressure;
* Hormone therapy in the period of 02 months prior to inclusion;
* Administration of any drug in the 02 weeks prior to inclusion;
* A history of autoimmune anemia or hereditary;
* research subjects with a history of chronic bleeding;
* research subjects with a history of acute bleeding in the last 30 days;
* History of sensitivity to biological products derived from mammals, albumin, or any component of the formulation;
* History of or current use at least 12 months of tobacco;
* Current or previous history (less than 12 months) of illicit drug use;
* previous therapy with erythropoietin;
* albumin below 3.5 g / dl or greater than 4.8 g / dL;
* Signs or clinical history of bone marrow aplasia;
* History of liver disease and clinical or laboratory;
* History of renal disease and clinical or laboratory.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-11; Primary Completion 2012-11 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic - rHuEPO concentration. | Before administration (Time 0 hour) and after time 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 11 hours, 12 hours, 13 hours, 18 hours, 24 hours, 36 hours, 48 hours, 72 hours, 96 hours and 120 hours administration.
  Will evaluated through the plasma rHuEPO dosage before and after drug administration.
Pharmacodynamics - Absolute Reticulocyte Count. | Before administration (Time 0 hour) and after Time 4 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours, 96 hours, 120 hours, 144 hours, 168 hours, 192 hours, 216 hours, 240 hours and 576 hours administration.
  Will evaluated through the absolute reticulocyte count at total blood.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Frederico, PI, Principal Investigator — LAL Clinica Pesquisa e Desenvolvimento Ltda
Locations (1):
- LAL Clínica Pesquisa e Desenvolvimento Ltda., Valinhos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
It is believed that after the data analysis and presentation to the National Commission on Research Ethics, all data will become public.